CLINICAL TRIAL: NCT06567340
Title: StratCare Trial 2: Evaluating the Clinical and Cost-effectiveness of AI-driven Stratified Care for Depression
Acronym: StratCare-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rotherham Doncaster and South Humber NHS Foundation Trust (Other Government)
Collaborators: University of Sheffield (Other); FSA Research Consulting Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 152958; 329457 (Other: IRAS); 153364 (Other Grant/Funding Number: NIHR HTA); NCT06728397 (obsolete NCT alias)
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Depression
Keywords: Software; Medical Devices; Mental Health; Anxiety; Psychotherapy; Cognitive Behavioural Therapy; Mood Disorders; Mental Health Services
MeSH Terms: conditions — Depression; Psychological Well-Being; Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Intervention Model Description: A pragmatic, single-blind, multi-site, parallel group cluster RCT. Cluster randomisation will be used to allocate Talking Therapies Teams and their patients to either intervention or usual care arms. In the experimental arm, treatment selection will be guided by an AI tool (StratCare app). In the USC arm, treatment will be selected following usual clinical practice and guidelines.
Who Masked: Participant, Outcomes Assessor
Masking Description: Trial statisticians will be blinded to allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- StratCare (Experimental): Treatment recommendation made by the StratCare-2 App using stratified care principles.
  Interventions: Device: StratCare
- Usual Stepped Care (No Intervention): Treatment recommendation made using usual stepped care principles.

INTERVENTIONS:
Device: StratCare — The StratCare app is a technology that collects data, processes inputs using a machine learning algorithm, and outputs a personalised treatment recommendation using automated decision rules. The inputs for the algorithm include patient-reported measures of depression, anxiety, functional impairment, personality traits, employment status and ethnic background. The algorithm calculates an expected prognosis (i.e., a probability of full remission of depression and anxiety symptoms after treatment), based on which patients are classified as standard (better expected prognosis) or complex cases. Standard cases are matched to low-intensity treatments and later have the option to move to high-intensity, whereas complex cases are matched directly to high-intensity treatments. In addition, the StratCare app is programmed to implement decision rules that ensure compliance with national clinical guidelines for the treatment allocation of patients with specific disorders.
  Arms: StratCare

SUMMARY:
Depression and anxiety are common mental health problems affecting around one in six adults. Treatments include therapy, telephone or group-based activities delivered by therapists. Treatment uses a "stepped care" model where most patients start with very brief treatments. If they remain unwell after this, they access longer and more intensive therapy. This model does not always work, as only one out of two patients fully recover.

The researchers have developed an artificial intelligence tool called "StratCare". It is designed to help health services to offer the best available treatment for each patient. StratCare is a computerised system that guides therapists on how to assess new patients. It asks a few questions about their symptoms, personality, and background. The system makes a recommendation about which treatment might be most effective for that person. This is either starting with brief therapy or starting with intensive therapy. The treatments are already used with depression in the National health Service (NHS). The patient can discuss with their therapist and decide whether to accept the recommendation. Otherwise, they can discuss trying other options. Previous research found that StratCare can help more people to recover from depression compared to the usual stepped care model.

The researchers will investigate if the StratCare tool works on a large scale in the NHS and if it helps patients in the long-term. The researchers will run a trial involving 1252 participants using NHS Talking Therapies services. Half will use the StratCare tool to make a treatment recommendation. The other half will follow the stepped care approach. The researchers will contact participants in the trial after 6, 12 and 18 months to see if their mood and quality of life has improved. The researchers will also interview therapists and participants to see what they think about treatment being guided by the StratCare tool.

Hypotheses:

* Stratified care will result in lower mean depression scores compared to usual stepped care (USC).
* Stratified care will result in a statistically significant higher proportion of cases with reliable and clinically significant improvement in depression symptoms, compared to USC.

Primary Outcome:

Depressive symptoms, as measured by change on the Patient Health Questionnaire (PHQ-9), at 12 months post-enrolment.

DETAILED DESCRIPTION:
Trial Design: A pragmatic, single-blind, multi-site, parallel group cluster Randomised Controlled Trial (RCT), with an internal pilot and stop/go criteria for progression to the full RCT. The researchers will recruit 1252 adult participants seeking treatment for common mental health problems who present with case-level depression symptoms on the Patient Health Questionnaire (PHQ-9) measure. They will be recruited from 16 services in the National Health Service (NHS) Talking Therapies programme across England.

Enrolment: Cluster randomisation will be used to allocate Talking Therapies Teams and their patients to either StratCare or Usual Stepped Care (USC) arms. Sites may have one or more Talking Therapies Teams participating in the trial.

After General Practitioner (GP) or self-referral for treatment, participants will undergo a standard clinical assessment by Talking Therapies clinicians, during which a treatment option will be selected. In the experimental arm, treatment selection will be guided by an Artificial Intelligence (AI) tool (StratCare app). In the USC arm, treatment will be selected following usual clinical practice and guidelines. Participants will then follow their selected treatment option.

NHS Trusts will be recruited through a Practice Research Network, NHS data service provider (PCMIS), and other means, attending to considerations of diversity and generalisability outlined in section seven. Within trusts, individual Talking Therapies teams will be recruited to participate in the trial. Randomisation will occur at team level rather than individual level, to reduce the risk of potential contamination from clinicians becoming aware of how the StratCare app makes treatment decisions.

Participants are adult patients seeking and eligible for treatment for common mental health problems in NHS Talking Therapies services. Patients who are eligible for treatment in the Talking Therapies service will be offered the opportunity to take part in the trial at the point of initial suitability assessment by the service, if seen by a team and clinician participating in StratCare-2.

Informed consent will be received verbally from participants during their initial assessment appointment with the treating Talking Therapies service. The StratCare App will guide clinicians through a brief and standardised script to provide information and seek verbal consent from patients who they assess in routine care. The researchers have chosen to obtain only verbal consent to minimize additional burden to make this viable within the constraints of routine care and due to the minimal risks posed by a new treatment selection method between two routinely delivered treatments.

A post consent 'opt-out' system is in place, so that once they have seen the full PIS, participants can withdraw from the trial shortly after consent and remove all their data. After the consent and assessment appointment, participants are sent a link to the participant information sheet (PIS), which provides further information on the study and how to opt out. If participants decide to withdraw their consent within a week of being sent the PIS, they will be classed as an opt-out, and all their information will be removed from trial records.

Treatment: Talking Therapies teams randomised to the experimental group will implement an AI-driven stratified care treatment pathway, where participants are matched to specific treatments based on their clinical and demographic features. Participants will complete a suitability assessment with a qualified assessing clinician. The assessing clinician will enter the required data from the clinical assessment, participant's previous treatment history and StratCare demographic items into the StratCare app which will give a treatment recommendation of low- or high-intensity treatment. The participant and clinician discuss the assessment outcome and make a joint decision about treatment based on the StratCare App recommendation. This joint decision does not have to follow the recommendation of the StratCare App. The decision will be recorded in the StratCare App and clinical records, and the participant will then proceed to the waiting list for the agreed treatment. If the decision does not follow the StratCare App recommendation, the reason for this will be recorded.

Talking Therapies teams randomised to the USC arm will complete a standard suitability assessment for the Talking Therapies service with a qualified assessing clinician. The StratCare App will be used by the assessing clinician to record the necessary data from the clinical assessment, the participant's previous treatment history and StratCare demographic items but the App will not be used to make a treatment recommendation. Treatment recommendation decisions will be made in the usual way, following stepped care principles - where most patients initially access low-intensity treatments and can subsequently access high-intensity treatments if the first step of care is unsuccessful. The participant and clinician discuss the assessment outcome and make a joint decision about treatment based on the clinician's recommendation. The decision will be recorded in clinical records, and the participant will then proceed to the waiting list for the agreed treatment.

Whichever group the participant is randomised to, they will still access the usual evidence-based interventions available in routine Talking Therapies services. These include low-intensity guided self-help, usually lasting up to eight sessions, and high-intensity psychological therapies which can last up to 20 sessions. These interventions will not be modified in any way, to preserve the integrity of routinely delivered care.

Assessing clinicians will be qualified Talking Therapies Psychological Wellbeing Practitioners (PWPs) or qualified Talking Therapies clinicians. Talking Therapies teams will have access and training (three hours) to use the StratCare technology described above, and study processes. Assessing clinicians will also be provided with bespoke Good Clinical Practice (GCP) training to cover the GCP principles required for their safe and ethical involvement in the trial, and an online portal for refresher training.

Data Collection: Data will be collected in five ways, depending on the stage of the trial, the type of data being collected, whether the participant is still being treated by the Talking Therapies service, and participant preference.

1. via direct entry into the StratCare App by the assessing clinician (baseline only).
2. as part of clinical care within the Talking Therapies service, collected by Talking Therapies staff. Data collected this way will be entered into the study database by study staff, or where available using an automated download from clinical records, transferred securely using an encrypted system to the study database.
3. via an online data collection system, self-reported.
4. via paper forms, self-reported.
5. via telephone or online video call, collected by study staff.

Data collection windows will be +/- one month of the target date. Where more than one data point exists within the data collection window, the data closest to the target date will be used. In exceptional circumstances where data does not exist within the data collection window, data within +/- three months can be used.

Whilst participants are in treatment, there will be routine collection of the PHQ-9 and GAD-7 measures. This data will not be used for the primary or secondary analyses, unless trial-collected data is missing for those time points. In this case, the routinely collected PHQ-9 or GAD-7 scores closest to the target dates, and within the data collection window, may be used.

Beyond the AI-guided treatment suggestion made by the StratCare App in the experimental arm, participant reported outcome data will not inform the clinical care of individual trial participants.

Safety: Further detail of adverse event reporting can be found within the protocol.

Statistical Analysis: The statistical analysis will follow intention-to-treat principles and CONSORT guidelines for Cluster RCTs and it will be pre-registered in an international register for controlled trials. The unit of inference for the StratCare-2 RCT, i.e., the quantity of interest that is to be estimated in a statistical analysis, is the effect of the intervention on a typical individual. Hence, the researchers are interested in the 'participant-average treatment effect', which answers the question 'How effective is the intervention for the average participant?'

Qualitative Sub-study: Semi-structured interviews with a purposive sample of clinicians and participants who took part in the trial will be conducted to carry out a process evaluation investigating implementation barriers, enablers, and factors affecting adherence to the AI-driven stratified care model. This will focus on aspects of "explainable" and "ethical" use of AI: (a) whether participants understand and accept AI-driven recommendations, and (b) whether there are situations where algorithmic recommendations are deemed clinically inappropriate by clinicians. Qualitative interviews will also capture information about participants' and clinicians' experiences of the shared decision-making process. Interviews will be analysed by the qualitative researcher using framework analysis. This will be informed by Sekhon's acceptability of healthcare interventions framework and Normalisation Process Theory, which can help identify whether interventions are likely to become embedded and integrated as part of routine practice or not.

Health Economic Analysis: An economic analysis will be conducted from the NHS and Personal Social Services perspective over the 18-month study time-horizon. A cost-utility analysis will use quality-adjusted life years (QALYs derived from the EuroQol-5D (EQ-5D) questionnaire, and tariff based on the United Kingdom public value set) as the measure of quality of life.

Process Evaluation: The researchers will collect fully pseudonymized clinical pathway and outcomes data for all participants to characterise the full treatment pathway for patients. Both quantitative (e.g., anonymised electronic health records data) and qualitative data will be used to undertake a thorough process evaluation of the logic model. Data on reach, dose and fidelity will be reported alongside qualitative findings on implementation, following guidelines for the process evaluation of complex interventions.

Evaluation of Generalisability: As StratCare-2 is embedded within each participating NHS Talking Therapies service where they all collect the nationally mandated outcome measures at each attended therapy session, the researchers will design a direct test of the generalisability of results obtained by trial participants with the wider population of attendees at these services. The researchers will seek permission to download data for each participating service/team for the time period two years preceding the start of each service/ teams' participation until the discharge of the final participant at a service/team.

Patient and Public Involvement and Engagement (PPIE): To ensure genuine, consistent partnership with patients and the public, two experienced PPIE Co-Leads will lead all PPIE input. The PPIE co-leads will conduct all the activities described in funder guidance (e.g., setting and refining the PPIE strategy as the project progresses). The researchers will run regular PPIE groups of up to 12 participants, comprising adult volunteers with lived experience of mental health problems and Talking Therapies services.

ELIGIBILITY:
Inclusion criteria:

* 18 years of age or older.
* Patients who consent to share their de-identified clinical records for research purposes.
* Patients assessed as eligible for psychological care in Talking Therapies based on clinical guidelines.
* Patients with case-level depression symptoms (PHQ-9 ≥ 10).

Exclusion Criteria:

• Those who are ineligible for treatment in Talking Therapies services according to standard treatment guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1252 (Estimated)
Dates: Start 2025-07-07 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms from enrolment, as measured by the Patient Health Questionnaire (PHQ-9) | 12 months post-enrolment.
  The PHQ-9 is a brief measure of depression symptoms, where each of 9 items is rated on a Likert scale from 0 to 3 representing symptom frequency in the last two weeks, yielding an overall severity score between 0 and 27. The cut-off ≥10 is recommended to screen for clinically significant depression symptoms, and a change of ≥6 points is indicative of statistically reliable change. The PHQ-9 has been extensively validated in primary care populations, with adequate sensitivity (88%) and specificity (88%) estimates for the detection of major depressive disorder using a cut-off score ≥10.

SECONDARY OUTCOMES:
Change in anxiety symptoms from enrolment, as measured by the Generalised Anxiety Disorder Questionnaire (GAD-7) | 6, 12 and 18 months post-enrolment.
  GAD-7 is a seven-item measure of common anxiety symptoms. Each item is scored on a 0-3 scale and these are summed to give an overall severity rating (range 0-21). The GAD-7 has been found to be a reliable screening tool for anxiety disorders such as generalised anxiety, social phobia, post-traumatic stress and panic disorder. A cut-off score ≥8 in this measure has been shown to detect an anxiety disorder with adequate sensitivity (77%) and specificity (82%).
Change in Quality of Life (to derive Quality Adjusted Life Years) from enrolment, as measured by the EQ-5D-5L | 6, 12 and 18 months post-enrolment.
  The 5-level EQ-5D (EQ-5D-5L) measure is commonly used to derive Quality Adjusted Life Years (QALYs) in healthcare research and to ensure that cost-effectiveness analyses are comparable to other studies and health technologies. Each of the five domain items is rated on a five-point scale from 'no problems' to 'extreme problems', giving a five-digit number describing the patients' health state. Patient responses will be converted into utility values using UK population tariff. Self-rated health is measured on a visual analogue scale from 0-100, with 100 being 'the best health you can imagine'. We will use the validated mapping function to derive utility values for the EQ-5D-5L questionnaire. QALYs will be calculated using the trapezoidal rule for calculating the area-under-the-curve, from baseline to the 18-month follow-up.
Change in Quality of Life from enrolment, as measured by the Recovering Quality of Life Scale 10 item version (ReQoL-10) | 6, 12 and 18 months post-enrolment.
  The ReQoL-10 was informed by contributions of >6,000 mental health service users. It has been developed specifically to assess quality of life in people with different mental health conditions and consists of 10 mental health questions and one physical health question. Each item is scored on a 0-4 scale and the 10 mental health scores are summed to give an overall score (range 0-40, 0 being poorest quality of life, 40 highest). A score of 24 or lower is considered as falling within the clinical range. An advantage of the ReQol-10 is that it captures a broad range of domains including meaningful activity, belonging and relationships, control and autonomy, hope, self-perception, well-being, and physical health.
Resource use across the trial duration, measured using an adapted Adult Service Use Schedule (AD-SUS) | 6, 12 and 18 months post-enrolment.
  Resource use data will include the following: (a) primary care consultations (e.g. appointments with physician and nurse practitioners); (b) Talking Therapies resource use (i.e. number of sessions at each step along the stepped care pathway - this is routinely collected for all Talking Therapies patients); (c) use of other mental health services (e.g. consultations with psychologists, psychiatrists, community psychiatric nurse); (d) hospital visits (e.g. emergency department visits, outpatient appointments and inpatient admissions); (e) use of medications; and (f) contacts with social care (e.g. social worker, home care worker, outreach worker).
Change in depressive symptoms from enrolment, as measured by the Patient Health Questionnaire (PHQ-9) | 6 and 18-months post enrolment.
  The PHQ-9 is a brief measure of depression symptoms, where each of 9 items is rated on a Likert scale from 0 to 3 representing symptom frequency in the last two weeks, yielding an overall severity score between 0 and 27. The cut-off ≥10 is recommended to screen for clinically significant depression symptoms, and a change of ≥6 points is indicative of statistically reliable change. The PHQ-9 has been extensively validated in primary care populations, with adequate sensitivity (88%) and specificity (88%) estimates for the detection of major depressive disorder using a cut-off score ≥10.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Delgadillo, Prof, Principal Investigator — University of Sheffield; Michael Barkham, Prof, Principal Investigator — University of Sheffield
Locations (1):
- Rotherham Doncaster and South Humber NHS Foundation Trust, Doncaster, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
StratCare-2 will share its data using a controlled access, data repository approach. After the closure of the trial, simplified, minimised, anonymised datasets will be made available within a recognised data repository. This will be within a 'controlled access system' (i.e. data access requires approval and compliance with a formal data sharing agreement), in line with United Kingdom Clinical Trials Network (UKCRN) )recommendations. A study-specific Data Sharing Plan will be agreed and approved by the sponsor, Trial Management Group (TMG), Trial Steering Committee (TSC) and Clinical Trials Research Unit (CTRU) Quality Assurance team prior to any data being deposited or shared. This will outline where data is stored, what is stored, and how access to it is requested, reviewed and approved.

REFERENCES:
- [Background] Bower P, Gilbody S. Stepped care in psychological therapies: access, effectiveness and efficiency. Narrative literature review. Br J Psychiatry. 2005 Jan;186:11-7. doi: 10.1192/bjp.186.1.11. PMID 15630118
- [Background] Delgadillo J, Moreea O, Lutz W. Different people respond differently to therapy: A demonstration using patient profiling and risk stratification. Behav Res Ther. 2016 Apr;79:15-22. doi: 10.1016/j.brat.2016.02.003. Epub 2016 Feb 23. PMID 26937855
- [Background] Delgadillo J, Lutz W. A Development Pathway Towards Precision Mental Health Care. JAMA Psychiatry. 2020 Sep 1;77(9):889-890. doi: 10.1001/jamapsychiatry.2020.1048. No abstract available. PMID 32459326
- [Background] Andrews G. Should depression be managed as a chronic disease? BMJ. 2001 Feb 17;322(7283):419-21. doi: 10.1136/bmj.322.7283.419. No abstract available. PMID 11179166
- [Background] Delgadillo J, Huey D, Bennett H, McMillan D. Case complexity as a guide for psychological treatment selection. J Consult Clin Psychol. 2017 Sep;85(9):835-853. doi: 10.1037/ccp0000231. PMID 28857592
- [Background] Goddard E, Wingrove J, Moran P. The impact of comorbid personality difficulties on response to IAPT treatment for depression and anxiety. Behav Res Ther. 2015 Oct;73:1-7. doi: 10.1016/j.brat.2015.07.006. Epub 2015 Jul 16. PMID 26226089
- [Background] Clark DM. Realizing the Mass Public Benefit of Evidence-Based Psychological Therapies: The IAPT Program. Annu Rev Clin Psychol. 2018 May 7;14:159-183. doi: 10.1146/annurev-clinpsy-050817-084833. Epub 2018 Jan 19. PMID 29350997
- [Background] Delgadillo J, Ali S, Fleck K, Agnew C, Southgate A, Parkhouse L, Cohen ZD, DeRubeis RJ, Barkham M. Stratified Care vs Stepped Care for Depression: A Cluster Randomized Clinical Trial. JAMA Psychiatry. 2022 Feb 1;79(2):101-108. doi: 10.1001/jamapsychiatry.2021.3539. PMID 34878526
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Moran P, Leese M, Lee T, Walters P, Thornicroft G, Mann A. Standardised Assessment of Personality - Abbreviated Scale (SAPAS): preliminary validation of a brief screen for personality disorder. Br J Psychiatry. 2003 Sep;183:228-32. doi: 10.1192/bjp.183.3.228. PMID 12948996
- [Background] Hingorani AD, Windt DA, Riley RD, Abrams K, Moons KG, Steyerberg EW, Schroter S, Sauerbrei W, Altman DG, Hemingway H; PROGRESS Group. Prognosis research strategy (PROGRESS) 4: stratified medicine research. BMJ. 2013 Feb 5;346:e5793. doi: 10.1136/bmj.e5793. PMID 23386361
- [Background] Hussain JA, White IR, Johnson MJ, Byrne A, Preston NJ, Haines A, Seddon K, Peters TJ. Development of guidelines to reduce, handle and report missing data in palliative care trials: A multi-stakeholder modified nominal group technique. Palliat Med. 2022 Jan;36(1):59-70. doi: 10.1177/02692163211065597. Epub 2022 Jan 17. PMID 35034529
- [Background] Keetharuth AD, Brazier J, Connell J, Bjorner JB, Carlton J, Taylor Buck E, Ricketts T, McKendrick K, Browne J, Croudace T, Barkham M. Recovering Quality of Life (ReQoL): a new generic self-reported outcome measure for use with people experiencing mental health difficulties. Br J Psychiatry. 2018 Jan;212(1):42-49. doi: 10.1192/bjp.2017.10. PMID 29433611
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] van Hout B, Janssen MF, Feng YS, Kohlmann T, Busschbach J, Golicki D, Lloyd A, Scalone L, Kind P, Pickard AS. Interim scoring for the EQ-5D-5L: mapping the EQ-5D-5L to EQ-5D-3L value sets. Value Health. 2012 Jul-Aug;15(5):708-15. doi: 10.1016/j.jval.2012.02.008. Epub 2012 May 24. PMID 22867780
- [Background] Byford S, Barrett B, Metrebian N, Groshkova T, Cary M, Charles V, Lintzeris N, Strang J. Cost-effectiveness of injectable opioid treatment v. oral methadone for chronic heroin addiction. Br J Psychiatry. 2013 Nov;203(5):341-9. doi: 10.1192/bjp.bp.112.111583. Epub 2013 Sep 12. PMID 24029536
- [Background] Offorha BC, Walters SJ, Jacques RM. Statistical analysis of publicly funded cluster randomised controlled trials: a review of the National Institute for Health Research Journals Library. Trials. 2022 Feb 4;23(1):115. doi: 10.1186/s13063-022-06025-1. PMID 35120567
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- [Background] Clark TP, Kahan BC, Phillips A, White I, Carpenter JR. Estimands: bringing clarity and focus to research questions in clinical trials. BMJ Open. 2022 Jan 3;12(1):e052953. doi: 10.1136/bmjopen-2021-052953. PMID 34980616
- [Background] Lawrance R, Degtyarev E, Griffiths P, Trask P, Lau H, D'Alessio D, Griebsch I, Wallenstein G, Cocks K, Rufibach K. What is an estimand & how does it relate to quantifying the effect of treatment on patient-reported quality of life outcomes in clinical trials? J Patient Rep Outcomes. 2020 Aug 24;4(1):68. doi: 10.1186/s41687-020-00218-5. PMID 32833083
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Murray E, Treweek S, Pope C, MacFarlane A, Ballini L, Dowrick C, Finch T, Kennedy A, Mair F, O'Donnell C, Ong BN, Rapley T, Rogers A, May C. Normalisation process theory: a framework for developing, evaluating and implementing complex interventions. BMC Med. 2010 Oct 20;8:63. doi: 10.1186/1741-7015-8-63. PMID 20961442
- [Background] Manca A, Hawkins N, Sculpher MJ. Estimating mean QALYs in trial-based cost-effectiveness analysis: the importance of controlling for baseline utility. Health Econ. 2005 May;14(5):487-96. doi: 10.1002/hec.944. PMID 15497198
- [Background] Briggs AH, Wonderling DE, Mooney CZ. Pulling cost-effectiveness analysis up by its bootstraps: a non-parametric approach to confidence interval estimation. Health Econ. 1997 Jul-Aug;6(4):327-40. doi: 10.1002/(sici)1099-1050(199707)6:43.0.co;2-w. PMID 9285227
- [Background] Fenwick E, Byford S. A guide to cost-effectiveness acceptability curves. Br J Psychiatry. 2005 Aug;187:106-8. doi: 10.1192/bjp.187.2.106. PMID 16055820
- [Background] Husereau D, Drummond M, Augustovski F, de Bekker-Grob E, Briggs AH, Carswell C, Caulley L, Chaiyakunapruk N, Greenberg D, Loder E, Mauskopf J, Mullins CD, Petrou S, Pwu RF, Staniszewska S; CHEERS 2022 ISPOR Good Research Practices Task Force. Consolidated Health Economic Evaluation Reporting Standards 2022 (CHEERS 2022) Statement: Updated Reporting Guidance for Health Economic Evaluations. Value Health. 2022 Jan;25(1):3-9. doi: 10.1016/j.jval.2021.11.1351. PMID 35031096
- [Background] Relton C, Torgerson D, O'Cathain A, Nicholl J. Rethinking pragmatic randomised controlled trials: introducing the "cohort multiple randomised controlled trial" design. BMJ. 2010 Mar 19;340:c1066. doi: 10.1136/bmj.c1066. No abstract available. PMID 20304934
- [Background] Tudur Smith C, Hopkins C, Sydes MR, Woolfall K, Clarke M, Murray G, Williamson P. How should individual participant data (IPD) from publicly funded clinical trials be shared? BMC Med. 2015 Dec 17;13:298. doi: 10.1186/s12916-015-0532-z. PMID 26675031
- [Background] Staniszewska S, Brett J, Simera I, Seers K, Mockford C, Goodlad S, Altman DG, Moher D, Barber R, Denegri S, Entwistle A, Littlejohns P, Morris C, Suleman R, Thomas V, Tysall C. GRIPP2 reporting checklists: tools to improve reporting of patient and public involvement in research. BMJ. 2017 Aug 2;358:j3453. doi: 10.1136/bmj.j3453. PMID 28768629
- [Background] Cohen ZD, DeRubeis RJ. Treatment Selection in Depression. Annu Rev Clin Psychol. 2018 May 7;14:209-236. doi: 10.1146/annurev-clinpsy-050817-084746. Epub 2018 Mar 1. PMID 29494258
- [Background] Saunders R, Cape J, Fearon P, Pilling S. Predicting treatment outcome in psychological treatment services by identifying latent profiles of patients. J Affect Disord. 2016 Jun;197:107-15. doi: 10.1016/j.jad.2016.03.011. Epub 2016 Mar 8. PMID 26991365
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- See also: National Institute of Health Research (NIHR) Research Funding Award StratCare-2 — https://www.fundingawards.nihr.ac.uk/award/NIHR153364